CLINICAL TRIAL: NCT02841020
Title: The Effect of Pre-treatment Biopsy for Non-neoplastic Renal Disease vs no Biopsy on Estimated Glomerular Filtration Rate in Patients With Small Renal Mass: a Single-center, Single-blinded, Randomized, Parallel Group Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for study fell through
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Noah Schenkman, MD, Associate Professor of Urology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 19081
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2017-11

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control SOC (No Intervention): Standard of care is followed
- Experimental additional biopsy (Experimental): Additional biopsy
  Interventions: Procedure: Additional biopsy

INTERVENTIONS:
Procedure: Additional biopsy — • Patients in the experimental group receive the additional biopsy for non-neoplastic disease during the same procedure before the biopsy of the renal mass (with potential for direct benefit to the patient by revealing non-neoplastic renal disease).
  Arms: Experimental additional biopsy

SUMMARY:
The purpose of this study is to determine if biopsy for non-neoplastic renal disease for patients with a small renal mass results in greater postoperative renal function than the current standard of care (no additional biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater
* Scheduled for renal biopsy as part of clinical care
* Diagnosis of small renal mass (< 4cm) based on imaging (CT, MRI, Ultrasound, or other)
* Patient must provide written, informed consent for study procedures before randomization
* Renal mass must be primarily solid (as opposed to cystic) in nature

Exclusion Criteria:

* Patients less than 18 years of age
* Patients who are prisoners
* Women who are pregnant-self reported
* Patients with Bosniak 3 or 4 cystic renal masses
* Patients with history of renal transplantation
* Patients with eGFR less than 30-based on review of clinical labs
* Patients on dialysis
* Patients with bleeding disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
difference in change in glomerular filtration rate (GFR) | 6 months